CLINICAL TRIAL: NCT01294722
Title: The Prevalence of Out-patients With Rheumatoid Arthritis Fulfilling the Indication for Anti-tumor Necrosis Factor(TNFa) Therapy in General Hospital Setting in Korea: a Multi-center, Non-interventional, Observational Study
Brief Title: A Study to Determine the Number of Participants With Rheumatoid Arthritis (RA) Who Meet the Requirements for Treatment With Anti-Tumor Necrosis Factor α (TNFα) in a General Hospital Setting in Korea
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100769; REMICADEARA4015 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; anti-TNF α
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study to estimate the proportion of patients diagnosed with RA visiting a medical internist in a general hospital in Korea who are candidates for anti-TNF α therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA
* Visiting a medical internist in a study site during the study period on out patient basis
* Able to give written informed consent voluntarily Exclusion Criteria: None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with diagnosis of RA visiting an internist as an outpatient
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Actual)
Dates: Start 2011-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of anti-TNF α agent candidates fulfilling the reimbursement guideline of Korea government in total out-patients with RA | Baseline
Number of anti-TNF α agent candidates based on the clinical judgement in total out- patients with RA | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (1):
- Seoul, South Korea